CLINICAL TRIAL: NCT01524653
Title: Impact of Rosuvastatin on Risk Markers of Venous Thromboembolism During Systemic Therapy for Advanced Cancer
Brief Title: Detecting the Impact of Statin Therapy On Lowering Risk of Venous Thrombo-Embolic Events (DISOLVE)
Acronym: DISOLVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Steven Ades, Assistant Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VCC 1110
Record Dates: First submitted 2012-01-20; First posted 2012-02-02 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Neoplasms
Keywords: VTE; DVT; Chemo; Metastatic; Advanced; Systemic therapy; statin; biomarkers
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Neoplasms; Neoplasm Metastasis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin First, Placebo Last (Experimental): This arm will receive rosuvastatin during the first treatment period followed by placebo in the second treatment period after washout.
  Interventions: Drug: Rosuvastatin; Drug: Placebo
- Placebo First, Rosuvastatin Last (Experimental): This arm will receive placebo during the first treatment period followed by rosuvastatin in the second treatment period after washout.
  Interventions: Drug: Rosuvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — 20 mg po od
  Other Names: Crestor
Drug: Placebo — 20 mg po od

SUMMARY:
Patients with cancer have a high risk of developing venous blood clots or thromboembolism (VTE). In an effort to target patients at highest risk of VTE for thromboprophylaxis (protective treatment for blood clots), numerous studies have identified serum biomarkers for risk of future VTE. There is also increasing evidence pointing to a prophylactic effect of statin therapy on the risk of developing VTE in high-risk populations including patients with advanced cancer. The purpose of this research study is to find out whether treatment with rosuvastatin (the study drug) reduces the risk of VTE in patients with cancer receiving chemotherapy. This study is specifically investigating the impact of rosuvastatin therapy on serum biomarkers (D-dimer and others) that indicate a risk for VTE, as well as safety and tolerance of rosuvastatin therapy in this population.

This is a phase II randomized crossover study with two 3-4 week treatment periods during which all enrolled patients will receive 20 mg of rosuvastatin once a day by mouth or a matching placebo tablet. Approximately two tablespoons of blood will be collected for biomarker analysis at the beginning and end of each treatment period. After the first treatment period there will be a 3-5 week break where subjects will undergo a washout. Following this washout period every subject will "crossover" or begin taking the alternative therapy so everyone enrolled will receive the study drug either during the first or the second treatment period. Biomarker levels will be analyzed in both treatment periods and compared to baseline, with every patient acting as their own control.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years old with locally-advanced or metastatic cancers who are about to start or are already receiving any systemic chemotherapy or targeted therapy.
* Estimated overall survival of ≥ 6 months
* Anticipated duration of therapy ≥ 9 weeks (if 3-week cycle) or ≥ 12 weeks (if 2 or 4-week cycle). Systemic therapy is allowed to change if necessary, or to terminate, during this period

Exclusion Criteria:

* Antithrombotic therapy including warfarin, dabigatran, low molecular weight heparin or unfractionated heparin. Patients taking aspirin may participate in this study.
* Anti-angiogenic therapy with thalidomide or lenalidomide. Patients receiving bevacizumab may participate in this study.
* Patients starting hormonal therapy exclusively, such as SERM or aromatase inhibitor therapy for breast cancer, or androgen-ablative therapy for prostate cancer.
* Statin use within 3 months prior to enrolment
* Adjuvant therapy in patients who have already received curative-intent local therapy (surgery or radiotherapy). Patients with glioblastoma starting adjuvant chemotherapy are an exception given the high likelihood of residual disease and risk of VTE in this population.
* Asian descent as assessed by history. If either of the participant's parents is Asian (peoples of East, Southeast, and South Asia), a patient will be excluded due to slower metabolism of the drug and concerns regarding toxicity at the 20 mg dose level.
* Urinary creatinine clearance of less than 40 ml/min based on reported MDRD GFR, present in FAHC metabolic profile reports, during the 14 day screening period.
* AST or ALT elevation of greater than 3X upper limit of normal, during the 14 day screening period.
* Patients with a known history of statin intolerance that was accompanied by severe adverse reaction.
* Patients who are currently participating in another clinical trial involving an investigational medication if there is a known or suspected drug interaction with rosuvastatin or the statin class, or if the investigational agent is known or suspected to be associated with a significantly increased risk of thrombosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-03; Primary Completion 2016-07-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
To determine if rosuvastatin therapy reduces the risk of VTE in patients with cancer receiving chemotherapy, as measured by a decrease in D-dimer level with treatment compared to placebo | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)

SECONDARY OUTCOMES:
To investigate the impact of rosuvastatin therapy on other established biomarkers of VTE risk in cancer patients receiving chemotherapy as measured by the change in Factor VIII | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)
To investigate the impact of rosuvastatin therapy on other established biomarkers of VTE risk in cancer patients receiving chemotherapy as measured by the change in soluble P-selectin | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)
To investigate the impact of rosuvastatin therapy on other established biomarkers of VTE risk in cancer patients receiving chemotherapy as measured by the change in C-reactive protein | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)
To investigate the impact of rosuvastatin therapy on other established biomarkers of VTE risk in cancer patients receiving chemotherapy as measured by the change in Peak thrombin generation | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)
Adverse Events (CTCAE v4) associated with rosuvastatin therapy | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)
  Liver toxicity and rhabdomyolysis
Venous thromboembolism | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)
  Clinical signs of venous thromboembolism
To investigate the impact of rosuvastatin therapy on other established biomarkers of VTE risk in cancer patients receiving chemotherapy as measured by the change in Plasminogen activator inhibitor-1 activity | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)
To investigate the impact of rosuvastatin therapy on other established biomarkers of VTE risk in cancer patients receiving chemotherapy as measured by the change in Plasminogen activator inhibitor-1 protein concentration | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)
To investigate the impact of rosuvastatin therapy on other established biomarkers of VTE risk in cancer patients receiving chemotherapy as measured by the change in tissue factor | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)
To investigate the impact of rosuvastatin therapy on other established biomarkers of VTE risk in cancer patients receiving chemotherapy as measured by the change in Factor XIa | baseline, 3-4 weeks, 6-9 weeks, 9-13 weeks (ranges depending one treatment period lengths set for each patient at enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ades, MD, MSc, Principal Investigator — University of Vermont
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States

REFERENCES:
- See also: Vermont Cancer Center — http://www.vermontcancer.org/